CLINICAL TRIAL: NCT03028675
Title: pH-weighted MRI in Multiple Sclerosis: A Surrogate Marker of Tissue Metabolic Stress
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01434
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Multiple Sclerosis
  Interventions: Other: MRI Scan
- Healthy Volunteer: 10 age-matched control volunteers
  Interventions: Other: MRI Scan

INTERVENTIONS:
Other: MRI Scan — MRI scans will consist of a 1-hour brain scan for both patients and controls.

SUMMARY:
Twenty subjects (10 patients and 10 age-matched control volunteers) will be recruited for this study. MRI scans will take place on a 3T MRI Scanner (Skyra or Prisma, Siemens Medical Solutions) located at The NYU Center for Biomedical Imaging. MRI scans will consist of a 1-hour brain scan for both patients and controls. In the first 6 months of the study, investigators will develop and test a uMT-based APT imaging for brain tissue pH measurement and use a hypercapnia paradigm to validate the tissue pH changes between breathing room air and 5% CO2 (by increasing tissue acidity) inhalation. With implementation of hypercapnia MRI, pH-weighted imaging will be validated for its robustness and reproducibility.

DETAILED DESCRIPTION:
The contrast agent (Gd-DTPA, Gadavist) will be injected intravenously (IV) in the arm (patients only). The IV will be inserted by qualified medical professional at CBI. This contrast agent will be standard dose in accordance with its FDA approved labeling and dosing. Controls will NOT be administered the contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female non-MS control volunteers

Exclusion Criteria:

* Medically unstable or with cardiac, pulmonary, hematological, renal, or hepatic dysfunction.
* Current or past DSM-IV diagnosis of major depression, bipolar and psychotic disorders.
* Contraindications for MRI, including
* Intracranial clips
* Metal implants
* External metallic devices/objects/clips within 10mm of the head
* Suspected or confirmed metal in the eyes (history of welding or similar activity)
* Claustrophobia
* Cardiac pacemaker or pacing wires
* Pregnancy - Pregnancy tests will be offered to women of childbearing age at no cost to the subject
* History of moderate to severe head injury, stroke, and seizures.
* Alcoholism or drug dependency.
* Renal or liver disease as this may cause concerns related to Gd-DTPA contrast agent.

  * Allergy to the contrast agent Gadolinium
  * Relapses or steroid therapy in patient at or in the month preceding the study
  * Patients only

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with relapse-remitting multiple sclerosis from NYU Langone Health and age-matched healthy volunteers recruiting using previous database of volunteers
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
pH measurements | 20 Minutes
  The pH will be estimated based on the calibration methods of quantification of exchange as a function of saturation time (QUEST)32 and its ratiometric analysis (QUESTRA) 33.

CONTACTS AND LOCATIONS:
Overall Officials: Yulin Ge, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States